CLINICAL TRIAL: NCT01242501
Title: Randomized Trial of a Brief HIV Risk Reduction Counseling Intervention for Sexually Transmitted Infections Clinic Patients in Cape Town, South Africa
Brief Title: Brief HIV Prevention Counseling for STI Patients in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H05-113
Record Dates: First submitted 2010-11-15; First posted 2010-11-17 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Sexually Transmitted Infections
Keywords: Prevention; Counseling; Behavioral interventions; HIV risk reduction
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: 3 Group RCT
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 60 Min. Risk Reduction Counseling (Experimental): Single 60 min Social Cognitive Theory-based counseling session delivered in STI clinic setting in Cape Town South Africa. Includes educational, motivational, and sexual risk reduction skills components delivered in a single face-to-face counseling session.
  Interventions: Behavioral: 60 Minute HIV/STI risk reduction counseling.Single 60 min Social Cognitive Theory-based counseling.
- 20-min single session education (Active Comparator): Single brief HIV/STI education only session for men and women receiving sexually transmitted infection clinic services in South Africa. Includes only brief educational information on sexual risks for HIV infection in a single face-to-face counseling session.
  Interventions: Behavioral: 20-Min education session

INTERVENTIONS:
Behavioral: 60 Minute HIV/STI risk reduction counseling.Single 60 min Social Cognitive Theory-based counseling. — Single session risk reduction counseling delivered in STI clinic settings in South Africa.
  Arms: 60 Min. Risk Reduction Counseling
Behavioral: 20-Min education session — Patients receive a single 20 min education session for STI/HIV informationSingle brief HIV/STI education only session for men and women receiving sexually transmitted infection clinic services in South Africa. Includes only brief educational information on sexual risks for HIV infection in a single face-to-face counseling session.
  Arms: 20-min single session education

SUMMARY:
This is a randomized trial to test a brief single session risk reduction counseling intervention on HIV and STI behavioral outcomes in Cape Town South Africa.

DETAILED DESCRIPTION:
This 5 year study will conduct a randomized clinical trial of a gender and culturally tailored theory-based behavioral risk reduction intervention for men and women who are receiving sexually transmitted infection (STI) diagnostic and treatment services from STI treatment providers in South Africa. As many as one in five South Africans is HIV positive and there are an estimated 1,500 new HIV infections in South Africa each day. The experimental intervention in this study was developed by South African and US investigators and pilot tested in South Africa. The intervention is grounded in the experience of South African health service provider, empirical research on AIDS-related stigmas, and elements of a social cognitive theory of health behavior change. The intervention consists of a single 60-minute risk reduction counseling session delivered within the context of STI services. Participants will be STI clinic patients over age 18 that have been treated for a previous STI. Participants will be baseline assessed and randomized to receive either (a) the 60 min theory-based and culturally tailored risk reduction intervention or (b) a time and contact matched standard of care HIV and health education session. Participants will be followed for 12 months post intervention. Assessments will be conducted using computer assisted interviews (ACASI). The randomized trial will determine the efficacy of the risk reduction intervention for South African men and women receiving STI clinic services. Outcome analyses will include differences between conditions on new STI diagnoses over 12 months. We will also test the mediating effects of attitudes and beliefs on intervention outcomes. Results of this research will therefore test a clinic-based HIV prevention intervention model that is urgently needed in South Africa.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* STI clinic patient diagnosed with an STI at current visit

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Chart abstracted sexually transmitted infections | 12 month aggregate
  STI clinic chart abstracted diagnoses over 12 month observation period.

SECONDARY OUTCOMES:
Sexual behavior change | 3-month intervals
  Computer assisted interview behavioral assessments of sexual risk and risk reduction.

CONTACTS AND LOCATIONS:
Overall Officials: Seth Kalichman, Ph.D., Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

REFERENCES:
- [Result] Kalichman SC, Cain D, Eaton L, Jooste S, Simbayi LC. Randomized clinical trial of brief risk reduction counseling for sexually transmitted infection clinic patients in Cape Town, South Africa. Am J Public Health. 2011 Sep;101(9):e9-e17. doi: 10.2105/AJPH.2011.300236. Epub 2011 Jul 21. PMID 21778486